CLINICAL TRIAL: NCT05240456
Title: Safety and Efficacy Beta 3 Agonists in Treatment of Non-neurogenic Voiding Dysfunction in Children, a Randomized Clinical Trial
Brief Title: Beta 3 Agonists in Treatment of Non-neurogenic Voiding Dysfunction in Children
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Islam Mansour, Principal invistigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS.21.09.1680
Record Dates: First submitted 2021-12-11; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Voiding Disorders; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Adrenergic beta-3 Receptor Agonists; Cholinergic Antagonists; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This arm will receive standard behavioral therapy plus Mirabegron with adjusted-dose regimen (25-50 mg), patients of 20-40 kg will receive 25-50 mg once a day; patients >40 kg will receive 50 mg once a day, for three months.
  Interventions: Drug: Beta3-Agonists, Adrenergic
- Control (Active Comparator): This arm will receive will receive standard behavioral therapy plus Solifenacin with a daily dosage of (2.5-10 mg/kg), for three months.
  Interventions: Drug: Anticholinergic drug, Solifenacin

INTERVENTIONS:
Drug: Beta3-Agonists, Adrenergic — The beta 3 agonist ,Mirabegron, has been shown to be effective for the treatment of OAB in adults through relaxation of bladder wall, with few side effects. This intervention aims to evaluate its efficacy and safety for children with non-neurogenic voiding dysfunction.
  Other Names: Standard behavioral Urotherapy
  Arms: Intervention
Drug: Anticholinergic drug, Solifenacin — Anticholinergic drugs are widely used to treat overactive bladder by relaxation of bladder wall smooth muscles.
  Other Names: Standard behavioral Urotherapy
  Arms: Control

SUMMARY:
A randomized clinical study to evaluate the safety and efficacy of using the Beta 3 agonist drug (Mirabegron) combined with standard behavioral therapy in comparison to using the anticholinergic drug (Solifenacin) combined with behavioral therapy, for children with non-neurogenic voiding dysfunction refractory to behavioral therapy alone, using improvement of dysfunctional voiding symptom score as a primary measurement of efficacy.

DETAILED DESCRIPTION:
The study aims to evaluate the beta 3 agonist drug (Mirabegron) as regard its safety and efficacy when used in children with non neurogenic voiding dysfunction, including children suffering from frequency, urgency, urgency incontinence and hesitancy who do not have neurological disease explaining these symptoms and who failed behavioral urotherapy.

The patients will be randomly allocated into two groups, one will receive standard behavioral therapy plus Mirabegron, the other will receive standard behavioral therapy plus the anticholinergic drug Solifenacin for three months. Patients will be assessed initially and after three months using:

* Medical and voiding history (bladder voiding diary, Dysfunctional voiding symptom score (DVSS) , Bristol Stool Scale)
* Dysfunctional voiding symptom score (DVSS) , Bristol Stool Scale
* Urine analysis and mid-stream urine culture.
* Uroflowmetry.
* Pelvic US and post-void residual urine (PVR).

ELIGIBILITY:
Inclusion Criteria:

* Children with non-neurogenic voiding dysfunction predominantly filling phase dysfunctions or OAB, refractory to behavioral therapy as a primary monotherapy, with dysfunctional voiding symptom score of ≥6 for females and ≥9 for males, between the age of 5 & 18 years old.

Exclusion Criteria:

* Neurogenic or anatomical bladder problems.
* Patients with contraindications to Beta 3 agonists or anticholinergic drugs.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Beta 3 agonist drug (Mirabegron) in improving symptoms of children with voiding dysfunction using dysfunctional voiding scoring system as a primary measure. | 6 months.
  To evaluate the efficacy of using the Beta 3 agonist drug (Mirabegron) combined with standard behavioral therapy in comparison to using the anticholinergic drug (Solifenacin) combined with behavioral therapy, for children with non-neurogenic voiding dysfunction refractory to behavioral therapy alone, using improvement of dysfunctional voiding symptom score as a primary measurement of efficacy. This score consists of 10 voiding dysfunction parameters that are assigned scores of 0 to 3 according to prevalence, and possible total scores ranging from 0 to 30. The higher the score, the more severe the symptoms of voiding dysfunction. The documented cutoff score for voiding dysfunction is 6 and 9 for females and males respectively.

SECONDARY OUTCOMES:
To evaluate the side effects of the beta 3 agonist drug (Mirabegron) in children. | 6 months
  This is planned to assess side effects and safety profile of the beta 3 agonist (Mirabegron) on children (5-18 years) from Egypt.
To validate an Arabic version of the Dysfunctional Voiding Scoring System as the documented cutoff score for voiding dysfunction is 6 and 9 for females and males respectively. | 6 months
  The investigators are planning to translate an Arabic version of the Dysfunctional Voiding Scoring System to use it to assess improvement of symptoms and patient recorded outcomes for Egyptian children before and after receiving Mirabegron.
To evaluate correlation between bladder ultrasound findings and severity of patients' symptoms. (normally it is less than 3 mm) | 6 months
  The investigators are planning to assess Ultrasound measurement of bladder wall thickness as an indicator of severity of patients' symptoms and whether there is bladder wall hypertrophy corresponding to severity of symptoms and whether the bladder wall thickness decreases with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Islam Mansour, Mb ChB, Principal Investigator — Mansoura University

IPD SHARING:
Plan to Share IPD: No